CLINICAL TRIAL: NCT04794621
Title: Electroceutical Dressing Technology Against Wound Microbial Biofilm Infection
Brief Title: Electroceutical Dressing Technology (EDT) Against Wound Microbial Biofilm Infection
Acronym: EDT BioFilm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Sashwati Roy, Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012285504
Record Dates: First submitted 2021-02-25; First posted 2021-03-12 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Wound Heal
Keywords: surgical wounds; infected wounds
MeSH Terms: conditions — Surgical Wound; Wound Infection

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: to avoid bias, the personnel performing the biofilm analysis (Primary outcome) will be blinded towards the study groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care Only (No Intervention): This will be group 1
- SOC and PED-10 +Procellera (Experimental): In group 2, in addition to SoC, the patients will apply the EDThi dressing (PED-10) on the wound(s) for the first 3 weeks following enrollment followed by Procellera® or EDTlo for additional 3 weeks. The use of dressings will be discontinued anytime if complete wound closure is achieved.
  Interventions: Device: Electroceutical Dressing Technology-EDThi; Device: Adding EDTlo (Procellera®) for 3 weeks after use of EDThi

INTERVENTIONS:
Device: Electroceutical Dressing Technology-EDThi — Use of EDThi for 3 weeks post enrollment
  Other Names: Standard Of Care
  Arms: SOC and PED-10 +Procellera
Device: Adding EDTlo (Procellera®) for 3 weeks after use of EDThi — Use of EDTlo (Procellera®) for additional 3 weeks
  Arms: SOC and PED-10 +Procellera

SUMMARY:
There are currently limited treatments available that show anti-biofilm efficacy for wound infection management Biofilms account for over 80% of infections and approximately 65% of nosocomial infections caused by microorganisms in the developed world involve biofilms. There clearly is a need for cost effective, highly stable, easily obtained biofilm targeted strategies for treatment of chronic wound biofilm infections.

The information generated from this project has the potential of providing considerable benefits to wound care by determining the efficacy of EDT dressing in managing wound biofilm infection and efficacy in wound healing and closure. Such knowledge could help therapeutic strategies and could provide information for future clinical studies to further understanding -of EDT wound dressings.

DETAILED DESCRIPTION:
This is a randomized open-label clinical study to test the efficacy of the treatment protocol using an optimized EDThi & EDTlo sequential approach in infected or high risk of infection burn/trauma/surgery chronic wounds against biofilm infection. This trial will determine the efficacy of EDT dressing against wound biofilm infection. subjects will be randomized to one of the two groups: 1) standard of care (SoC) only and 2) SoC + EDT dressing treatment. In group 2, in addition to SoC, the patients will apply the EDThi dressing (PED-10) on the wound(s) for the first 3 weeks following enrollment followed by Procellera® for additional 3 weeks. The use of dressings will be discontinued anytime if complete wound closure is achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 years and older
2. subjects willing and able to provide informed consent
3. patients with infected chronic trauma or surgical wounds
4. wound(s) must be able to be covered by the EDT dressing
5. All patients, with wounds below the knee, must have wound tissue oxygenation adequate to support wound healing per provider discretion, this may be defined by one or more of the following perfusion values within 6 months on enrollment: peri-wound transcutaneous oxygen measurements ≥ 25 mmHg (TCOM),Ankle Brachial Index (ABI) >0.7, or a Toe pressure (TP) > 40 mmHg, If none of these tests were performed during standard of care, then a trained study team member may obtain a TCOM measurement after the patient has consented and before they are enrolled. If there are multiple perfusion values that conflict, then a physician will review and determine if they are eligible for enrollment. If a patient has had a recent re-vascularization, the patient may be enrolled once adequate perfusion has been verified.
6. Subjects must be able to read and understand English.

Exclusion Criteria:

1. Individuals who are deemed unable to understand the procedures, risks and benefits of the study, ie. Informed consent will be excluded
2. Pregnant women
3. Prisoners
4. Wound tissue not available for analysis
5. Patient with known sensitivity or allergic reaction to zinc or silver
6. Current active diagnosis of Osteomyelitis at the target wound site, that is untreated, based on clinical diagnosis per EMR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Response to the use of EDT treatment in prevention of wound biofilm infection | 6 weeks
  Impact of EDT treatment in prevention of incidence of wound biofilm infection

SECONDARY OUTCOMES:
rate of wound closure 6 weeks post-treatment as compared to baseline | 6 weeks
  rate of wound closure 6 weeks post-treatment as compared to baseline
wound microbiome in SoC and SoC+ EDT treatment. | 3 weeks
  presence of microbiome in standard of care with and w/o treatment
Percent of patients with response to EDT treatment on week 6 as compared to SoC only group | 6 weeks
  Percent of patients showing treatment response on week 6 comparing SOC group to ntervention group

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, PhD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Eskenazi Health, Indianapolis, Indiana
  - Richard L. Roudebush VA Medical Center, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT04794621/ICF_000.pdf